CLINICAL TRIAL: NCT06212661
Title: Migraine Medication Effects on Urinary Symptoms
Status: Enrolling by invitation | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Howard Goldman, MD, Principal investigator / Professor and Vice Chair (Quality and Patient Safety) Glickman Urologic and Kidney Institute, The Cleveland Clinic
Other Study IDs: 23-1101
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Overactive Bladder; Bladder Pain Syndrome; Migraine Disorders; Overactive Bladder Syndrome; Overactive Detrusor; Migraine; Interstitial Cystitis
MeSH Terms: conditions — Urinary Bladder, Overactive; Cystitis, Interstitial; Migraine Disorders | interventions — ubrogepant; rimegepant sulfate; atogepant; eptinezumab; fremanezumab; erenumab; galcanezumab; Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CGRP inhibitor: * Ubrogepant (Ubrelvy™)
  * Rimegepant (Nurtec®)
  * Atogepant (Qulipta™)
  * Eptinezumab (Vyepti®)
  * Fremanezumab (Ajovy®)
  * Galcanezumab (Emgality®)
  * Erenumab (Aimovig®) dosage and duration according to provider's clinical decision.
  Interventions: Drug: Ubrogepant; Drug: Rimegepant; Drug: Atogepant; Drug: Eptinezumab; Drug: Fremanezumab; Drug: Galcanezumab; Drug: Erenumab
- BoNTA extracranial muscle injections: Botolinum toxin A (Botox) Injection into extracranial muscles to treat migraine. Dosage and duration according to provider's clinical decision
  Interventions: Drug: Botulinum toxin A

INTERVENTIONS:
Drug: Ubrogepant — Ubrogepant (Ubrelvy™), oral, dosage at discretion of clinical provider, for treatment of migraine headaches.
  Other Names: Ubrelvy
  Groups: CGRP inhibitor
Drug: Rimegepant — Rimegepant (Nurtec®), oral, dosage at discretion of clinical provider, for treatment of migraine headaches.
  Other Names: Nurtec
  Groups: CGRP inhibitor
Drug: Atogepant — Atogepant (Qulipta™), oral, dosage at discretion of clinical provider, for treatment of migraine headaches.
  Other Names: Qulipta
  Groups: CGRP inhibitor
Drug: Eptinezumab — Eptinezumab (Vyepti®) injection, dosage at discretion of clinical provider, for treatment of migraine headaches.
  Other Names: Vyepti
  Groups: CGRP inhibitor
Drug: Fremanezumab — Fremanezumab (Ajovy®) injection, dosage at discretion of clinical provider, for treatment of migraine headaches.
  Other Names: Ajovy
  Groups: CGRP inhibitor
Drug: Galcanezumab — Galcanezumab (Emgality®) injection, dosage at discretion of clinical provider, for treatment of migraine headaches.
  Other Names: Emgality
  Groups: CGRP inhibitor
Drug: Erenumab — Erenumab (Aimovig®) injection, dosage at discretion of clinical provider, for treatment of migraine headaches.
  Other Names: Aimovig
  Groups: CGRP inhibitor
Drug: Botulinum toxin A — Botolinum toxin A (Botox) injections into extracranial muscles, dosage at discretion of clinical provider, for treatment of migraines.
  Other Names: Botox
  Groups: BoNTA extracranial muscle injections

SUMMARY:
A prospective observational cohort trial to study the effects of CGRP inhibitors (CGRPi) on lower urinary tract symptoms (LUTS) and bladder/pelvic pain. Candidates for either CGRPi or an alternative therapy for refractory migraines (OnabotulinumtoxinA (BoNTA) extracranial muscle injections) with baseline LUTS will be recruited. The investigators will assess LUTS and pelvic pain using validated symptom and quality-of-life questionnaires, pretreatment and at 3 months post-treatment follow-up, comparing change in symptoms based on treatment received.

DETAILED DESCRIPTION:
Common urinary urgency syndromes may be related to over-activation of bladder afferent pathways involving CGRP signaling. CGRP (calcitonin gene related protein) is a neurotransmitter in afferent pathways also involved in central nociception and hypersensitization. CGRP-targeted therapies, approved for migraine treatment, have the potential to alleviate lower urinary tract symptoms, but these possible effects have not been studied in humans.

This is a prospective observational cohort trial to study the effects of CGRP inhibitors (CGRPi) on lower urinary tract symptoms (LUTS) and bladder/pelvic pain. Candidates for either CGRPi or an alternative therapy for refractory migraines (OnabotulinumtoxinA (BoNTA) extracranial muscle injections) with baseline LUTS will be recruited. The investigators will assess LUTS and pelvic pain using validated symptom and quality-of-life questionnaires, pretreatment and at 3 months post-treatment follow-up, comparing change in symptoms based on treatment received.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients > 18 years
* Refractory migraine, planned treatment with either:
* CGRP inhibitors, including:

  * CGRP small molecule receptor antagonists ("gepants"): Ubrogepant, Rimegepant, Atogepant.
  * CGRP monoclonal antibodies: Eptinezumab, Fremanezumab, Galcanezumab.
  * CGRP receptor monoclonal antibodies: Erenumab.
* BoNTA extracranial muscle injections
* Any of the following symptoms during the last month:

  * Urinating too often (frequency).
  * Having a sudden urge to urinate that's difficult to hold back (urgency).
  * Having a sudden urge to urinate and urine leaking before you make it to the toilet (urge incontinence).

Exclusion Criteria:

* Age < 18 years
* CGRP treatment within the last 12 months or BoNTA (head / bladder) last 6 months.
* Patient (or medical decision-maker) unable to provide informed consent or unable to answer questionnaire.
* Unable to urinate, eg: post cystectomy, indwelling catheter, on intermittent self catheterization, ESRD w/ anuria.
* Prior bladder BoNTA in last 12 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients age 18 years or over, presenting to the neurology outpatient clinics for treatment of refractory migraine with either CGRP inhibitors or Botulinum toxin extracranial muscle injections, and with at least 1 urinary storage-phase symptom in the past month.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
changes in OAB symptoms | 3 months
  To prospectively compare changes in OAB symptoms after beginning CGRP inhibitor treatment for migraine, with changes after beginning local BoNTA injections for migraine as controls.
  OAB symptom change will be measured using the International Consultation on Incontinence Questionnaire (ICIQ) - Female Lower Urinary Tract Symptoms (FLUTS). ICIQ-FLUTS questionnaire composite OAB score, including urgency, frequency, nocturia and urge incontinence domains (range: 0-16, higher scores indicate worse symptoms). Differences of 2-4 points with a standard deviation of 3-4 points were reported as significant in the literature.

SECONDARY OUTCOMES:
changes in bladder pain symptoms | 3 months
  To prospectively compare changes in bladder pain symptoms after beginning CGRP inhibitor treatment for migraine, with changes after beginning local BoNTA injections for migraine as controls.
  Bladder / pelvic pain symptom change will be measured using the Female Genitourinary Pain Index (GUPI). The score ranges from 0 to 39, quality of life question score from 0 to 6, and higher scores indicate worse symptoms.
rates of LUTS and LUTS-related quality of life (QoL) in patients with chronic refractory migraine. | 3 months
  To assess rates of LUTS (Lower Urinary Tract Symptoms) and LUTS-related quality of life (QoL) in patients with chronic refractory migraine.
  LUTS will be assessed using the International Consultation on Incontinence Questionnaire (ICIQ) - Female Lower Urinary Tract Symptoms (FLUTS). This questionnaire has 12 symptoms questions scored 0 to 4, overall questionnaire score is 0 to 48 points, and higher scores indicate worse symptoms.
  Bladder / pelvic pain symptoms will be measured using the Female Genitourinary Pain Index (GUPI). The score ranges from 0 to 39, higher scores indicate worse symptoms.
  LUTS-related quality of life question, adopted from the international prostate symptom score (IPSS) or American Urological Association symptom index (AUASI), is scored 0 to 6 and a higher score indicated worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Howard B Goldman, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
no plan to share with other researchers